CLINICAL TRIAL: NCT05351684
Title: Effect of Dolutegravir Intensification on Blood and Tissue Latent HIV-1 Reservoirs and on Residual Viremia Despite ART
Brief Title: Effect of Dolutegravir Intensification on HIV-1 Reservoirs
Acronym: EDIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Gilles Darcis, Principal Investigator, University of Liege
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-228
Record Dates: First submitted 2019-10-24; First posted 2022-04-28 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intensified (Experimental): Group of patients whose treatment will be intensified with an additional 50mg of dolutegravir on top of regular treatment (Triumeq: ABC/3TC/DTG).
  Interventions: Drug: Dolutegravir 50 MG
- Control (No Intervention): Group of patients without modification of baseline treatment (Triumeq: ABC/3TC/DTG).

INTERVENTIONS:
Drug: Dolutegravir 50 MG — already included in arm/group descriptions.
  Arms: Intensified

SUMMARY:
Persistent HIV viremia occurs in most ART-treated patients and could arise from reactivation of viral expression from latently-infected cells that constitute the viral latent reservoir (LR) and/or residual ongoing viral replication during cART, for instance in anatomical compartment where drug penetration is sub-optimal.

The question of the sources of persistent viremia is of the utmost importance. If ongoing viral replication occurs, it could induce deleterious consequences on reservoirs size and immune activation.We propose to better characterize the role ongoing viral replication to HIV persistence under ART by undertaking a treatment intensification trial with high-dose dolutegravir. Tissue/blood samples and replication-competent reservoir measurements will be included as outcomes as well as immune activation markers.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected adults receiving cART for at least 3 years
* Undetectable viral for at least 3 years
* DTG/3TC/ABC as cART regimen in the previous 6 months.
* CD4 counts higher than 200 cells per μL

Exclusion Criteria:

* active hepatitis C or B
* unstable liver disease
* renal impairment (estimated glomerular filtration rate <50 mL per min),
* gastrointestinal disorders that would affect the absorption of study treatment
* current use of drugs with significant interactions with dolutegravir
* current use of drugs with an impact on inflammation such as steroids.
* hospitalization for acute illness within the previous 8 weeks
* Pregnancy or breastfeeding.
* Anal or rectal lesions impeding rectal biopsies
* Decreased platelets count or coagulation disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-08-28 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of treatment intensification at the level of total and replication-competent reservoir (RCR) in blood and in tissues. | 3 months
  Measurements of blood and tissue HIV reservoir

SECONDARY OUTCOMES:
To evaluate the impact of DTG treatment intensification on residual viremia | 3 months
  Measurement of HIV viremia at the single copy level
To evaluate the impact of DTG treatment intensification on immune activation | 3 months
  Measurement of T cell activation markers
To investigate the correlation between blood and tissues HIV reservoir | 3 months
  Measurement of blood and tissue HIV reservoir
To correlate the concentration of DTG with residual viremia and impact on HIV reservoir | 3 months
  Measurement of DTG blood concentration
To evaluate the impact of DTG treatment intensification on inflammation | 3 months
  Measurement on inflammatory markers in blood

CONTACTS AND LOCATIONS:
Locations (1):
- Liège university hospital, Liège, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fombellida-Lopez C, Valaitiene A, Winchester L, Maes N, Dellot P, Vanwinge C, Ladang A, Cavalier E, Susin F, Vaira D, Hayette MP, Reenaers C, Moutschen M, Fletcher CV, Pasternak AO, Darcis G. Doubling dolutegravir dosage reduces the viral reservoir in ART-treated people with HIV. Elife. 2026 Jan 23;14:RP106931. doi: 10.7554/eLife.106931. PMID 41575190